CLINICAL TRIAL: NCT00997438
Title: Defining the Anti-inflammatory Role of Lipoic Acid in Multiple Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Portland VA Medical Center (U.S. Federal Agency)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Daniel Carr, Research Career Scientist, Portland VA Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5659; OHSU eIRB#5659 (Other: OHSU)
Record Dates: First submitted 2009-10-16; First posted 2009-10-19 (Estimated); Results first posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2016-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Thioctic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- MS - Secondary Progressive (Experimental): 1200 mg of Lipoic acid supplement
  Interventions: Dietary Supplement: Lipoic Acid
- MS - Relapsing Remitting (Experimental): 1200mg of Lipoic acid supplement
  Interventions: Dietary Supplement: Lipoic Acid
- Healthy Controls (Experimental): 1200 mg of Lipoic acid supplement
  Interventions: Dietary Supplement: Lipoic Acid

INTERVENTIONS:
Dietary Supplement: Lipoic Acid — 300 mg Lipoic acid tablets from Vital Nutrients

SUMMARY:
The purpose of this study is to learn about how the antioxidant, lipoic acid, works in the body and how it may help in the management of relapsing remitting and secondary progressive multiple sclerosis. This study will compare how subject's and healthy volunteers bodies absorb and break down the supplement. This information may help in developing new therapies.

DETAILED DESCRIPTION:
Subjects (healthy control, relapsing remitting MS and secondary progressive MS) will be recruited through patients of investigators at Portland VA Medical Center (PVAMC), Oregon Health & Science University (OHSU), and the community using flyers and word of mouth.

The following will occur during screening:

* Medical History Questionnaire to include questions about drug and alcohol use
* Self Administered Expanded Disability Status Scale (EDSS) Questionnaire (MS participants only)
* Vital Signs (heart rate, respiratory rate, blood pressure) will be measured and recorded
* Physical Exam (MS participants only unless necessary, based on the Medical History Questionnaire or vital signs, to ensure participant safety)
* Neurological Exam (MS participants only unless necessary, based on the Medical History Questionnaire or vital signs, to ensure participant safety)
* Weight
* Urine pregnancy test, if applicable
* Anemia testing by finger stick (approximately 1 drop)

The rest of the study involves

* Blood draws before lipoic acid is given, 1 hour, 2 hours, 3 hours, 4 hours, 24 and 48 hours after LA is given (3 ½ tablespoons)
* Subjects will receive breakfast before they take LA
* Subjects will take 4 - 300 mg capsules of lipoic acid (LA) for a total of 1200mg with about 1 cup of water

Blood will be processed to obtain plasma (from which lipoic acid concentrations will be measured) and PBMCs (from which cAMP and cytokines/chemokines will be measured).

ELIGIBILITY:
Inclusion/Exclusion criteria for MS subjects.

Inclusion criteria:

1. Adult at least 18 years of age able to provide informed consent
2. Currently diagnosed with relapsing remitting or secondary progressive MS

Exclusion criteria:

1. Self-reported current substance/alcohol abuse/dependence or sobriety for less than 90 days
2. History of traumatic brain injury as defined by a loss of consciousness of greater than 30 minutes
3. History of a medical condition associated with persisting cognitive problems or serious central nervous system dysfunction (e.g., brain tumor,dementia)
4. MS exacerbation within 30 days of study entry
5. Systemically administered corticosteroids within 30 days of study entry
6. Pregnant or breast-feeding
7. Anti-coagulant use such as Heparin, Coumadin, or Aspirin while enrolled in the study
8. Other significant health problem (e.g. active coronary heart disease, liver disease, pulmonary disease, diabetes mellitus) that might increase the risk of subject experiencing adverse events
9. Any condition which would make the subject, in the opinion of the investigator, unsuitable for the study
10. Anemia as indicated by a POC hemoglobin <12
11. Subjects of child bearing potential or subjects capable of causing pregnancy who are sexually active and unwilling to use effective contraceptive methods for the duration of the study

Inclusion/ Exclusion criteria for healthy controls.

Inclusion criteria:

1) Adult at least 18 years of age able to provide informed consent

Exclusion criteria:

1. Self-reported current substance/alcohol abuse/dependence or sobriety for less than 90 days
2. History of traumatic brain injury as defined by a loss of consciousness of greater than 30 minutes
3. History of a medical condition associated with persisting cognitive problems or serious central nervous system dysfunction (e.g., brain tumor,dementia)
4. Pregnant or breast-feeding
5. Anti-coagulant use such as Heparin, Coumadin, or Aspirin while enrolled in the study
6. Other significant health problem (e.g. active coronary heart disease, liver disease, pulmonary disease, diabetes mellitus) that might increase the risk of subject experiencing adverse events
7. Any condition which would make the subject, in the opinion of the investigator, unsuitable for the study
8. Anemia as indicated by a POC hemoglobin <12
9. Subjects of child bearing potential or subjects capable of causing pregnancy who are sexually active and unwilling to use effective contraceptive methods for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2010-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Carr, Ph.D, Principal Investigator — Portland VA Medical Center and Oregon Health & Science University
Locations (2):
- United States (2):
  - Oregon Health & Science University, Portland, Oregon
  - Portland VA Medical Center, Portland, Oregon

REFERENCES:
- [Derived] Fiedler SE, Yadav V, Kerns AR, Tsang C, Markwardt S, Kim E, Spain R, Bourdette D, Salinthone S. Lipoic Acid Stimulates cAMP Production in Healthy Control and Secondary Progressive MS Subjects. Mol Neurobiol. 2018 Jul;55(7):6037-6049. doi: 10.1007/s12035-017-0813-y. Epub 2017 Nov 15. PMID 29143287

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited at PVAMC and OHSU January 2012-December 2013 via fliers, word of mouth and MS clinic screening.
Groups:
- MS - Relapsing Remmitting: 1200mg of Lipoic acid supplement
  Lipoic Acid: 300 mg Lipoic acid tablets from Vital Nutrients
Period: Overall Study
Arm/Group | MS - Secondary Progressive | MS - Relapsing Remmitting | Healthy Controls
Started | 21 | 24 | 24
Completed | 16 | 21 | 20
Not Completed | 5 | 3 | 4
Not completed — Blood draw difficulty | 2 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Exclusion criteria at visit 1 | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MS - Secondary Progressive | MS - Relapsing Remmitting | Healthy Controls | Total
Number analyzed (Participants) | 16 | 21 | 20 | 57
Age, Continuous [Median (Full Range); unit: years] | 57.5 [39 to 69] | 51 [29 to 64] | 49.5 [26 to 65] | 54 [26 to 69]
Gender [Count of Participants; unit: Participants]
  Female | 10 | 14 | 12 | 36
  Male | 6 | 7 | 8 | 21

OUTCOME MEASURES:

1. Primary Outcome: Lipoic Acid Levels
Description: Plasma concentration of LA
Time Frame: 1 hour
Population: Plasma samples from one secondary progressive and one healthy control subject did not yield results for unknown reason(s).
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | MS - Secondary Progressive | MS - Relapsing Remmitting | Healthy Controls
Number analyzed (Participants) | 15 | 21 | 19
ng/mL | 1376.14 (359.41) | 1609.07 (312.47) | 1428.05 (330.02)

2. Primary Outcome: Lipoic Acid Levels
Description: Plasma concentration of LA
Time Frame: 2 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | MS - Secondary Progressive | MS - Relapsing Remmitting | Healthy Controls
Number analyzed (Participants) | 15 | 21 | 19
ng/mL | 1125.71 (291.40) | 1167.33 (205.02) | 1348 (205.91)

3. Primary Outcome: Lipoic Acid Levels
Description: Plasma concentration of LA
Time Frame: 3 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | MS - Secondary Progressive | MS - Relapsing Remmitting | Healthy Controls
Number analyzed (Participants) | 15 | 21 | 19
ng/mL | 667.86 (138.24) | 638.4 (114.41) | 793.89 (173.39)

4. Primary Outcome: Lipoic Acid Levels
Description: Plasma concentration of LA
Time Frame: 4 hours
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | MS - Secondary Progressive | MS - Relapsing Remmitting | Healthy Controls
Number analyzed (Participants) | 15 | 21 | 19
ng/mL | 268.6 (73.15) | 252.75 (33.85) | 394.1 (129.15)

5. Primary Outcome: Lipoic Acid Levels
Description: Plasma concentration of LA
Time Frame: 24 hour
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | MS - Secondary Progressive | MS - Relapsing Remmitting | Healthy Controls
Number analyzed (Participants) | 15 | 21 | 19
ng/mL | 0.78 (0.13) | 0.87 (0.05) | 0.78 (0.06)

6. Primary Outcome: Lipoic Acid Levels
Description: Plasma concentration of LA
Time Frame: 48 hour
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | MS - Secondary Progressive | MS - Relapsing Remmitting | Healthy Controls
Number analyzed (Participants) | 15 | 21 | 19
ng/mL | 0.55 (0.15) | 0.7 (0.05) | 0.57 (0.04)

7. Primary Outcome: cAMP Levels
Time Frame: 2 hours
Population: Useable PBMCs were not obtained from one healthy control and 2 relapsing remitting MS patients
Measure: Median (Inter-Quartile Range); unit: pmol cAMP/mg protein
Arm/Group | MS - Secondary Progressive | MS - Relapsing Remmitting | Healthy Controls
Number analyzed (Participants) | 16 | 19 | 19
pmol cAMP/mg protein | 75.9 [46 to 101.5] | 75.8 [56.8 to 113] | 96.6 [75.1 to 129.2]

8. Primary Outcome: cAMP Levels
Time Frame: 4 hours
Population: Useable PBMCs were not obtained from one healthy control and 2 relapsing remitting MS patients
Measure: Median (Inter-Quartile Range); unit: pmol cAMP/mg protein
Arm/Group | MS - Secondary Progressive | MS - Relapsing Remmitting | Healthy Controls
Number analyzed (Participants) | 16 | 19 | 19
pmol cAMP/mg protein | 72.6 [56.8 to 90.1] | 79.1 [59.9 to 108.2] | 103.5 [63 to 149.6]

9. Secondary Outcome: RANTES Levels
Time Frame: 24 hour
Population: Analyses were terminated when it became clear no consistent significant changes in RANTES were taking place.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | MS - Secondary Progressive | MS - Relapsing Remitting | Healthy Controls
Number analyzed (Participants) | 7 | 7 | 3
pg/mL | 47184.9 (15986.8) | 36281.4 (13713.1) | 76751.7 (44904.2)

10. Secondary Outcome: RANTES Levels
Time Frame: 48 hour
Population: Analyses were terminated when it became clear no consistent significant changes in RANTES were taking place.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | MS - Secondary Progressive | MS - Relapsing Remmitting | Healthy Controls
Number analyzed (Participants) | 7 | 7 | 3
pg/mL | 44905.8 (16659.6) | 42593.8 (13848.9) | 60578.5 (21878.8)

ADVERSE EVENTS:
Arm/Group | MS - Secondary Progressive | MS - Relapsing Remmitting | Healthy Controls
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/24 | 1/24
Other Adverse Events (participants affected / at risk) | 0/21 | 1/24 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MS - Secondary Progressive (N=21) | MS - Relapsing Remmitting (N=24) | Healthy Controls (N=24)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Subject fainted and suffered facial abrasions as a result. CT scan and neuro consult determined likely vasovagal reaction causing syncope.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MS - Secondary Progressive (N=21) | MS - Relapsing Remmitting (N=24) | Healthy Controls (N=24)
Exacerbation of pre-existing myelopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Subject indicated heat packs used prior to IV made have contributed to exacerbation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes